CLINICAL TRIAL: NCT06677996
Title: A Phase 1, Open-Label, Fixed Sequence, 1-way Crossover Study Examining the Effect of Itraconazole on the Pharmacokinetics, Safety and Tolerability After Varegacestat Single Dose Administration to Healthy Participants
Brief Title: A Phase 1 Study to Examine the Effects of Itraconazole After Single Dose Administration of Varegacestat (AL102) to Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immunome, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AL102-501
Record Dates: First submitted 2024-11-04; First posted 2024-11-07 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteer
Keywords: Drug-Drug Interaction; Pharmacokinetics
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Period 1: varegacestat administration for PK followed by Period 2: itraconazole and varegacestat administration for PK and DDI
  Interventions: Drug: varegacestat; Drug: Itraconazole (200 mg)

INTERVENTIONS:
Drug: varegacestat — Experimental intervention
Drug: Itraconazole (200 mg) — Intervention to evaluate DDI with experimental intervention

SUMMARY:
This is an open label, fixed sequence, 1-way crossover drug-drug interaction (DDI) study in healthy participants.

DETAILED DESCRIPTION:
This is a phase 1, open-label, fixed sequence, 1-way crossover study examining the effect of itraconazole on the pharmacokinetics, safety and tolerability after varegacestat single dose administration to healthy participants. This is a 2-period study. In period 1 a single dose of varegacestat will be administered with PK evaluated predose and up to 192 hours postdose. There will be a 14 -day washout between period 1 and period 2. In period 2, itraconzole will be administered once daily for 18 consecutive days. Beginning on Day 4 of Period 2 a single dose of varegacestat will be administered 30 minutes after itraconazole dosing. Blood samples for PK will be collected prior to varegacestat dosing and up to 744 hours post varegacestat dosing for varegacestat and its metabolite.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female (of non-childbearing potential only), 18 to 55 years of age, inclusive, at the screening visit.
* Medically healthy with no clinically significant medical history, physical examination, clinical laboratory profiles, vital signs, and ECGs, as deemed by the PI or designee

Exclusion Criteria:

* Mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
* History of any illness that, in the opinion of the PI or designee might confound the results of the study or poses an additional risk to the participant by their participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Effect of itraconazole on the PK of varegacestat in healthy participants. | Up to 5 weeks
  AUC0-t for varegacestat administered with and without itraconazole.
Effect of itraconazole on the PK of varegacestat in healthy participants. | Up to 5 weeks
  AUC0-inf for varegacestat administered with and without itraconazole.
Effect of itraconazole on the PK of varegacestat in healthy participants. | Up to 5 weeks
  Cmax for varegacestat administered with and without itraconazole.
Effect of itraconazole on the PK of varegacestat in healthy participants. | Up to 5 weeks
  Tmax for varegacestat administered with and without itraconazole.

SECONDARY OUTCOMES:
Safety and tolerability of varegacestat in the presence of itraconazole in healthy participants. | Up to 2 months
  Number of subjects who experience treatment-emergent adverse events (TEAEs)
Safety and tolerability of varegacestat in the presence of itraconazole in healthy participants. | Up to 2 months
  Number of subjects who experience abnormalities in clinical laboratory tests such as serum chemistry and hematology
Safety and tolerability of varegacestat in the presence of itraconazole in healthy participants. | Up to 2 months
  Number of subjects who experience 12-lead ECG abnormalities
Ctrough of itraconazole and hydroxy-itraconazole in combination with varegacestat in healthy participants. | Up to 5 weeks
  Ctrough. values on prior to dosing itraconazole

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Valentine, Principal Investigator — Celerion
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided